CLINICAL TRIAL: NCT06636084
Title: Vertical and Horizontal Mandibular Ridge Augmentation Techniques: A Randomized Controlled Clinical Trial Comparing Customized CAD/CAM Titanium Mesh Versus Reinforced Perforated PTFE Mesh
Brief Title: Vertical and Horizontal Mandibular Ridge Augmentation Techniques
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hom-Lay Wang, DDS, MSD, Ph D, Collegiate Professor of Periodontics and Professor of Dentistry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00262750
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Vertical Ridge Deficiency; Horizontal Ridge Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Customized CAD/CAM Titanium Mesh (Experimental): A customized CAD/CAM Titanium Mesh will be used to cover the bone graft
  Interventions: Procedure: Guided bone regeneration (GBR)
- Reinforced Perforated PTFE Mesh (RPM) (Active Comparator): A Reinforced Perforated PTFE Mesh membrane will be used to cover the bone graft
  Interventions: Procedure: Guided bone regeneration (GBR)

INTERVENTIONS:
Procedure: Guided bone regeneration (GBR) — A composite graft composed of a 50:50 proportion of autogenous bone and a demineralized bone mineral will be positioned around the bony defect or placed in the membrane, depending on the group randomization. The selected membrane will then be secured with screws to ensure a complete and stable coverage of the grafted area.

SUMMARY:
The purpose of this study is to compare alveolar ridge augmentation outcomes of two types of membranes for vertical and horizontal mandibular ridge augmentation: Customized CAD/CAM Titanium Mesh versus Reinforced Perforated PTFE Mesh (RPM).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Physical status according to the American Society of Anesthesiology (ASA) I or II, which includes patients who are systematically healthy or may suffer from mild to moderate, however well-controlled systemic diseases.
* Subjects having at least one free end saddle edentulous area of the posterior area of the mandible with moderate horizontal and vertical bone defects >≥3mm.
* Capacity to understand and accept the written conditions of the study.

Exclusion Criteria:

* Insufficient oral hygiene.
* Smoking habit of >10 cigarettes/day (self-reported).
* Abuse of alcohol or drugs.
* Pregnancy or individuals attempting to get pregnant (self-reported).
* Acute local or systemic infections.
* Uncontrolled diabetes or other metabolic disease.
* Severe hepatic or renal dysfunction.
* Autoimmune disorders.
* Patients who underwent radiotherapy in the last 5 years.
* Patients undergoing immunosuppressive therapy or who are immunocompromised.
* Any other contraindications for undergoing surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Ridge width changes in mm | 6 months
  Radiographic changes of the ridge width based on cone-beam computed tomography (CBCT) scan measurements
Ridge height changes in mm | 6 months
  Radiographic changes of the ridge width based on cone-beam computed tomography (CBCT) scan measurements

SECONDARY OUTCOMES:
Change in the mucosal thickness in mm | 6 months
  Change in the mucosal thickness due to the provided space from baseline to the surgical mesh removal using an ultrasound
Histological outcomes of the augmented bone | 6 months
  In terms of the amount of newly formed vital bone, residual graft particles, and connective tissue (CT)/other non-mineralized tissue components as a percentage
The volumetric bone gain of the grafted area in mm3 | 6 months
  Radiographic changes of bone volume based on cone-beam computed tomography (CBCT) scan measurements
Rate of complications | 6 months
  Percentage that had complications associated with each technique
Cost analysis | 6 months
  Difference in cost-effectiveness in dollars

CONTACTS AND LOCATIONS:
Overall Officials: Hom-Lay Wang, DDS MSD PhD, Principal Investigator — Department of Periodontics and Oral Medicine, University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States